CLINICAL TRIAL: NCT03125317
Title: Evaluating the Efficacy of Valsalva's Maneuver and Music Therapy on Peripheral Venous Cannulation Pain and Anxiety
Brief Title: Evaluating the Efficacy of Valsalva's Maneuver and Music Therapy on Peripheral Venous Cannulation
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: 17-KAEK-009
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-04

CONDITIONS: Cannulation,Pain
MeSH Terms: interventions — Music Therapy; Valsalva Maneuver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The music group: Participant will allow to listen any kind of music which they wish
  Interventions: Other: Music
- valsalva maneuver: participants will be asked to take a deep breath and exhale the air out in 15 seconds
  Interventions: Other: Valsalva maneuver
- The control group: no intervention
  Interventions: Other: control

INTERVENTIONS:
Other: Music — a kind of music which the participant likes will be listened using speakers
  Groups: The music group
Other: Valsalva maneuver — Participant will be asked to take a deep breath and exhale the air out in 15 seconds
  Groups: valsalva maneuver
Other: control — No intervention
  Groups: The control group

SUMMARY:
Evaluating the efficacy of Valsalva's maneuver and music therapy on peripheral venous cannulation pain and anxiety

DETAILED DESCRIPTION:
One hundred and fifty patients undergoing surgery were randomized to apply Valsalva's maneuver (the valsalva group) and music therapy(the music group) and a placebo (the control group) during peripheral venous cannulation (PVC). The patients' pain, anxiety, and satisfaction scores will be measured.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status 1 and 2, between the ages of 18 and 65, were scheduled for elective surgery

Exclusion Criteria:

* Patients with a history of anxiety disorders or hearing problem and preoperative pain.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that underwent surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-09 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | one month
  Pain intensity

SECONDARY OUTCOMES:
satisfaction scale | one month
  satisfaction level(worst,bad,none,good,better)

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tapar, Principal Investigator — Assistant professor
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided